CLINICAL TRIAL: NCT04167332
Title: Prospective Collection of Samples for Urothelial Cancer of Bladder
Acronym: ProCSUCaB
Status: Not yet recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); HistoGeneX (Unknown); MDx Health (Industry); Hospital Clinic of Barcelona (Other); Mosaiques Diagnostics and Therapeutics AG (Unknown); Biomedical Research Foundation, Academy of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: S59371
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Bladder Cancer
Keywords: Non-muscle-invasive bladder cancer; Progression; Recurrence; Registry; Prospective; Biomarker; Multi-omics
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Disease Progression; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood, urine, and bladder cancer tissue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NMIBC: Patients diagnosed with primary non-muscle-invasive bladder (NMIBC) cancer.
  No experimental intervention will be administered. NMIBC patients will be diagnosed, treated and followed up according to guidelines-based institutional routines.
  The clinical (demographic, operative and follow-up) and pathological data, and biosamples (blood, urine, bladder cancer tissue) of the patients will be collected in a completely anonymous way.

SUMMARY:
ProCSUCaB (Prospective Collection of Samples for Urothelial Cancer of Bladder) is a monocentric, non-interventional, prospective registry that will recruit newly diagnosed intermediate- and high-risk NMIBC patients in a tertiary center in Flanders.

DETAILED DESCRIPTION:
ProCSUCaB (Prospective Collection of Samples for Urothelial Cancer of Bladder) is a monocentric, non-interventional, prospective registry that will recruit newly diagnosed intermediate- and high-risk NMIBC patients in a tertiary center in Flanders.

Clinical data and biosamples (blood, urine, and BC tissue) will be collected from each patient at the initial diagnosis before the surgery and will be stored at -80 °C at the BioBank UZ Leuven after proper processing according to the protocol. High-throughput multi-omics (genomics, epigenomics, transcriptomics, proteomics, lipidomics, metabolomics) and immunohistopathology analyses will be performed on these samples.

Patients of both sex and aged ≥18 years, with a signal of clinical diagnosis of BC (symptoms and/or imaging), are eligible to participate in this study. Patients, who give their informed consent to collect their biological materials prior to surgery, will be included in the study after the histopathological diagnosis of the TURBT specimen shows an intermediate- or high-risk NMIBC. Only the data of the patients with a TCC, with the allowance of any variant histopathological subtype, will be analyzed.

All patients will be treated and followed up with the standard of care based on the recommendations of the EAU Guidelines according to their risk groups. All follow-ups will be scheduled for 5 years as most of the recurrences or progressions occur during this period.

To comply with local privacy laws, all demographic and clinical data (for initial diagnosis and following recurrences and/or progressions) will be prospectively stored in a specific database, which is implemented into the hospital's electronic patient file system, and protected by firewalls [24]. All patients will receive a study identification number, and names (or any other identifying data) will be removed from the collected biosamples; therefore, all -omics and pathology laboratories will not know the identity and clinical data of the patients. The correspondence between the study identification numbers and patient names will be kept by only the urology department in a secured database.

Blood, urine and BC tissue samples will be collected at the initial diagnosis for every patient. Blood and urine will be collected by the nurses in the inpatient department in the morning prior to TURBT. After processing by the dedicated personnel, they will be sent to the BioBank UZ Leuven, which has continuously monitored and alarmed freezers, robotic handling, and storage system, and has implemented the Standard Pre-analytical Code (SPREC).

Blood collection: In the morning prior to TURBT (between 07:00-11:00 am), blood will be taken from the patients into five separate tubes (4x 10 mL EDTA tubes for genomics, epigenomics, transcriptomics, and proteomics; 1x 6 mL EDTA tube for lipidomics and metabolomics). Collection date and time will be recorded in the 'Urine/Blood Sampling Form' by the nurse. All blood tubes will be inverted gently 10 times after blood collection. All EDTA tubes will immediately be put in the refrigerator at +4°C in upright position until centrifugation. All blood samples will be centrifuged within 4 hours of collection, and centrifuge date and time will be recorded in the 'Blood Processing and Storage Form'. After processing all blood samples according to the specific protocol of each analysis, all plasma/pellet/whole blood samples in cryovials will be sent to the BioBank UZ Leuven to be stored at -80 °C, and the date and time of the sample acceptance will also be recorded.

Urine collection: A total of 230 mL of mid-stream urine will be collected into five tubes from the second urine in the morning (between 07:00-11:00 am) before TURBT. The patient should be well hydrated. Collection date and time will be recorded in the 'Urine/Blood Sampling Form' by the nurse. The urine samples will immediately be stored at +4 °C in the refrigerator and processed within 2 hours after collection, and centrifuge date and time will be recorded in the 'Urine Processing and Storage Form'. After processing all urine samples according to the specific protocol of each analysis, all samples in cryovials will be sent to the BioBank UZ Leuven to be stored at -80 °C, and the date and time of the sample acceptance will also be recorded.

Tissue collection: During TURBT, if the tumor is large enough (>10 mm in diameter), a big chip that includes the tumor stalk will be cut with the resectoscope. The sample will be put in a cryovial, and sent to the BioBank immediately thereafter. The date and time of collection and acceptance will be recorded in the 'Tissue Sampling and Storage Form'. Cryosection will be performed from frozen samples by a uropathologist before -omics analyses to check for presence and area of intermediate- and high-risk NMIBC. After the uropathologist's report, frozen samples will be dissected to take parts enriched in tumor cells. The histopathological diagnosis of the patients will be made according to the hematoxylin-eosin (HE) staining of the slides from the formalin-fixed paraffin-embedded (FFPE) blocks, which will determine the ultimate inclusion of the intermediate- and high-risk NMIBC patients.

ELIGIBILITY:
Inclusion Criteria:

1. A signal of clinical diagnosis of bladder cancer (symptoms and/or imaging)
2. Giving informed consent to collect clinical data and biological materials prior to surgery
3. An approved pathological diagnosis of transitional cell carcinoma (TCC), with allowance of any variant histopathological subtype
4. An approved pathological diagnosis of non-muscle-invasive bladder cancer (NMIBC), with stages of carcinoma in situ (CIS), Ta (mucosa-confined) and T1 (submucosa infiltrating)

Exclusion Criteria:

1. Aged less than 18 years
2. Not giving or withdrawing informed consent
3. Tumor histopathological type other than TCC, such as adenocarcinoma, squamous cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sex and aged ≥18 years, with a signal of clinical diagnosis of bladder cancer (symptoms and/or imaging), who are willing to participate in this registry and who give their informed consent to collect their clinical data and biological materials prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Comprehensive multi-layered molecular characterization | In two years after completion of recruitment of planned number of patients
  Comprehensive multi-layered molecular characterization of intermediate- and high-risk NMIBC patients at the genomics, epigenomics, transcriptomics, proteomics, lipidomics, metabolomics, and immunohistopathology levels for disease recurrence and progression
Multi-biomarker panel for disease recurrence and progression | In two years after completion of recruitment of planned number of patients
  Identification of a multi-biomarker panel that integrates multidimensional and longitudinal data with harnessing the power of various -omics, systems biology approach, network analysis and predictive modeling for a better stratification of intermediate- and high-risk NMIBC patients into their risk of recurrence and progression
Multi-biomarker panel for response to BCG treatment | In two years after completion of recruitment of planned number of patients
  Identification of a multi-biomarker panel for molecular characterization of a patient subgroup who receive BCG treatment, identification of the pathways relevant to BCG treatment response, and stratification of those patients according to their predicted BCG response

CONTACTS AND LOCATIONS:
Overall Officials: Steven Joniau, MD, PhD, Principal Investigator — UZ Leuven; Frank Van Der Aa, MD, PhD, Principal Investigator — UZ Leuven

IPD SHARING:
Plan to Share IPD: Yes
Due to ethical restrictions, anonymized data are available upon request to the Steering Committee. Anonymized data and biosamples of the patients can be requested for conducting scientific studies. All requests will be evaluated by the Steering Committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of data and biosample collection.
Access Criteria: Upon request to the Steering Committee, and after request evaluated by the Steering Committee.

REFERENCES:
- [Derived] Akand M, Veys R, Ost D, Vander Eeckt K, Baekelandt F, Van Reusel R, Mattelaer P, Baekelandt L, Van Cleynenbreugel B, Joniau S, Van der Aa F. Cohort Profile: VZNKUL-NMIBC Quality Indicators Program: A Flemish Prospective Cohort to Evaluate the Quality Indicators in the Treatment of Non-Muscle-Invasive Bladder Cancer. Cancers (Basel). 2024 Oct 29;16(21):3653. doi: 10.3390/cancers16213653. PMID 39518090
- [Derived] Akand M, Muilwijk T, Van Cleynenbreugel B, Gevaert T, Joniau S, Van der Aa F. Prototol for the Prospective Sample Collection for Cancer of Bladder (ProCaB) Trial by the Cancer of the Bladder Leuven (CaBLe) Consortium. Eur Urol Open Sci. 2024 Oct 15;70:21-27. doi: 10.1016/j.euros.2024.09.006. eCollection 2024 Dec. PMID 39483518